CLINICAL TRIAL: NCT05588505
Title: Refinement and Testing of a New Cognitive-Behavioral Intervention to Treat Executive Dysfunction in College Students With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Cognitive-Behavioral Treatment of Attention Deficit Hyperactivity Disorder (ADHD) in College Students - Study 1
Acronym: ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: The City College of New York (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-0013
Record Dates: First submitted 2022-10-10; First posted 2022-10-20 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: In the first (open trial) phase of the study, all participants will receive group cognitive-behavioral therapy (CBT) for executive self-management skills, including time-management, organization, and planning. Students will be assessed on measures of ADHD symptoms and executive self-management skills before and at the conclusion of the 12-week treatment program. Each group session lasts 2 hours.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Behavioral Therapy delivered in a group format (Experimental): Participating students will be assessed before and after the 12-week group Cognitive-Behavioral intervention to ascertain their response to the treatment.
  Interventions: Behavioral: Cognitive-Behavioral Therapy Targeting Executive Dysfunction in College Students with ADHD

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy Targeting Executive Dysfunction in College Students with ADHD — The intervention is 12 weeks long, made up of one 2- hour session each week. These sessions are designed to help the participants develop strategies to improve their executive functioning skills including self- care, time management and organizational skills. These skills will also be applied to specific academic tasks such as note-taking during reading and lectures, organizing and conducting research, and writing papers.

SUMMARY:
College students with ADHD have significant difficulty effectively managing their time, organizing, planning, and completing their academic work. As a result, they typically have lower grade-point averages, more course failures and withdrawals, are more likely to be placed on academic probation and are less likely to graduate from college than students without ADHD. The purpose of this project is to refine and test a psychological intervention on campus to help students with ADHD develop these self-management skills so that they can be more successful in college and avoid these negative outcomes.

DETAILED DESCRIPTION:
Participants will be assessed pre- and post-intervention during interviews with the clinician-investigators and on several self-report questionnaires designed to assess their self-management of time, organization, and planning. Feedback of the results will be discussed with them, including any recommendations for further treatment.

ELIGIBILITY:
Inclusion Criteria:

* Student at The City College of New York
* Diagnosis of ADHD, Inattentive or Combined Subtype
* In good physical health

Exclusion Criteria:

* Actively abusing drugs or alcohol within the past 6 months
* Actively suicidal
* Diagnosis of borderline personality disorder
* Diagnosis of bipolar disorder
* Diagnosis of a psychotic disorder
* Neurological disorder (such as traumatic brain injury, brain tumor, Parkinson's)
* History of childhood abuse or trauma or psychiatric condition that prevents clear
* confirmation of the presence of ADHD in childhood
* Any other acute psychiatric condition (e.g. acute panic disorder, severe depression) with treatment needs that take precedence over ADHD.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Adult Investigator Symptom Rating Scale (AISRS) at six months | Change from Baseline AISRS at six months
  The AISRS is a structured diagnostic Interview, administered by one of the study investigators to assess for Adult ADHD. Scores are reported on a scale from 0 to 27, with higher score being worse.
Change from Baseline Behavior Rating Scale of Executive Function - Adult Version (BRIEF-A) at six months | Change from Baseline BRIEF-A at 6 months
  The Meta-Cognitive Index of the BRIEF-A will be used to measure change in executive functions, including time-management, organization, and planning. Scores are reported as percentiles from 0 to 99 with a higher score being worse.
Change from Baseline Learning and Study Strategies Inventory (LASSI) at six months | Change from Baseline LASSI at 6 months
  The LASSI is a self-rating scale that measures student awareness and use of learning and study strategies on 10 scales related to skill, will, and self-regulation. Scores are reported as percentiles from 0 to 99 with a higher score being better.

CONTACTS AND LOCATIONS:
Overall Officials: Mary V. Solanto, Ph.D., Principal Investigator — Northwell Health; Anthony Rostain, M.D., Principal Investigator — Cooper School of Medicine at Rowan University
Locations (1):
- City College of New York, New York, New York, United States